CLINICAL TRIAL: NCT06069284
Title: Prognostic Significance of Acute Change in Liver and Splenic Stiffness in Patients of Acute on Chronic Liver Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-ACLF-12
Record Dates: First submitted 2023-09-15; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Acute on Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Acute-on-chronic liver failure (ACLF) is a syndrome associated with a high short- term mortality. Early identification of patients at high risk is important to determine emergency for transplantation and prioritize the need for intensive care unit. Unbalanced systemic inflammatory response is closely associated with mortality in ACLF patients. This systemic inflammatory response in ACLF increases liver and splenic stiffness stiffnes, which can be detected by transient elastography.

Very few studies have been done in past evaluating liver and splenic stiffness as prognostic tool in patients of ACLF. These studies have taken only single value of liver and splenic stiffness as prognostic tool. No follow up study have yet been done assessing acute change in liver and splenic stiffness in ACLF. In this study, we hypothesize that acute change in liver and splenic stiffness at 7th & 14 th day predicts outcome in ACLF patients. With this study, we aim to evaluate whether acute changes in liver and splenic stiffness at 7th & 14th day predicts outcome at 3 months in patients of ACLF.

DETAILED DESCRIPTION:
Study Design 1 year prospective cohort study Hypothesis: We hypothesize that acute change in liver and splenic stiffness at 7th & 14 th day predicts outcome in ACLF patients

Aim and Objective - Primary objective: To study the change in liver and splenic stiffness values at day 7 from baseline at day 1 between those with or without transplant free survival at Day 90.

Secondary objectives:

1) To study the change in liver and splenic stiffness values at day 14 from baseline at day 1 between those with or without transplant free survival at Day 90.

1. To evaluate association of baseline and change in liver and splenic stiffness with different etiologies of ACLF
2. To evaluate association of baseline liver and splenic stiffness with grade of esophageal varices in ACLF patients.
3. To evaluate association of baseline and change in liver and splenic stiffness with pattern of organ failures.
4. To evaluate association of changes in level of biochemical inflammatory markers with change in liver and splenic stiffness.
5. To evaluate association of baseline liver and splenic stiffness with severity of ACLF by AARC-ACLF score,CLIF-C-ACLF score, MELD-Na and CTP at presentation.
6. To evaluate change in liver and splenic stiffness with change in AARC-ACLF score and CLIF-C-ACLF score.

Methodology:

Study population All the consecutive patients of ACLF admitted in Hepatology wards will be evaluated for inclusion criteria

Study design: Prospective cohort study

Study period: 1 year after IEC approval.

Sample size: Consecutive patients of ACLF from approval of study to 12 months. 200 patients will be enrolled in our study

Intervention: None

Monitoring and assessment: All enrolled patients will undergo detailed evaluation by thorough history, clinical examination and relevant laboratory investigations. Patients will be graded as per AARC score grade I (5-7), II (8-10), III (11-15). CBC /NLR, KFT, LFT, PT/INR at baseline and alternate day, till discharge or death/Liver transplantation. TNF alpha, IL-6, CRP, ferritin, lactate at day 1, day 7 and day 14. AARC-ACLF score and CLIF-C-ACLF score at day 1, day 7 and day 14.USG abdomen and hepatic vein, porto-splenic doppler study will be performed in all cases and triple phase CT of abdomen when there will be suspicion of HCC. Fibroscan of liver and spleen at day 1, day 7 and day 14.UGI endoscopy will be performed within 7 days.

Initial Liver and Splenic stiffness and follow-up tests (Liver and splenic stiffness, TNF-alpha, IL-6) will be done free of cost.

STATISTICAL ANALYSIS:

Baseline data will be expressed as a proportion(%), the continuous data will be presented as mean+-SD OR mean ± SD or median ( IQR).

To compare between the groups, either, Student's t-test/ Mann Whitney test will be applied, as appropriate.

The categorical data will be analysed using χ2test or Fisher's exact test. The change between pre- and post-values will be analysed using paired t-test or McNemar test.

Significance defined as 2-tailed p-value of less than 0.05. Survival curves will be represented using Kaplan-Meier method.

ITT/ Per protocol analysis will be carried out for final result assessment. The data will be entered in Microsoft excel format and to be analysed using SPSS version 22 (IBM corp Ltd.; Armonk NY, USA).

Adverse effects: NA

ELIGIBILITY:
Inclusion Criteria:

1. Patients of ACLF as per APASL criteria between 18 to 70 years of age
2. Patient and attendants willing to give informed consent

Exclusion Criteria:

1. Age <18 years and > 70 years
2. Survival less than 7 days
3. Cirrhosis with prior decompensation
4. Grade 3 ascites
5. Hepatic encephalopathy grade III &IV
6. HCC/SOL >2cm in liver
7. Patient with congestive heart failure
8. Patient with extrahepatic cholestasis
9. Portal vein thrombosis
10. BMI >30 kg/m2
11. Prior variceal endotherapy or ongoing beta blocker treatment for varices
12. Pregnant and lactating women
13. Patient with cardiac pacemaker
14. Critically ill patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the consecutive patients of ACLF admitted in Hepatology wards will be evaluated for inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-25 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Acute changes in liver and splenic stiffness on day 7 in patients of ACLF predicts liver transplant free survival at 3 months. | 3 months

SECONDARY OUTCOMES:
Acute changes in liver and splenic stiffness on day 14 in patients of ACLF predicts liver transplant free survival at 3 months | 3 months
Association of baseline and change in liver and splenic stiffness with etiology of ACLF | Day 14
Association of baseline liver and splenic stiffness with severity of ACLF by AARC-ACLF score, at presentation | Day 1
Association of baseline liver and splenic stiffness with severity of ACLF by CLIF-C-ACLF score, at presentation | Day 1
Association of baseline liver and splenic stiffness with severity of ACLF by MELD-Na at presentation | Day 1
Association of baseline liver and splenic stiffness with severity of ACLF by CTP at presentation | Day 1
Association of baseline liver and splenic stiffness with grade of esophageal varices in ACLF patients | 1-7 days
Association of baseline and change in liver and splenic stiffness with pattern of organ failures. | Day 14
Association of changes in level of biochemical inflammatory markers with change in liver and splenic stiffness. | Day 14
Association of change in liver and splenic stiffness with change in AARC-ACLF score. | Day 14
Association of change in liver and splenic stiffness with change in CLIF-C-ACLF score. | Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: No